CLINICAL TRIAL: NCT04062682
Title: Impact of Healthy Diet on Metabolic Health in Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Horizon 2020 - European Commission (Other)
Responsible Party: Principal Investigator, Fawzi Kadi, Professor, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017/511
Record Dates: First submitted 2019-08-14; First posted 2019-08-20 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Healthy Aging; Metabolic Syndrome; Diet, Healthy
MeSH Terms: conditions — Metabolic Syndrome | interventions — Diet, Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controls (No Intervention): No changes in dietary habits
- Healthy Diet (Experimental): Changes in dietary habits only
  Interventions: Behavioral: Healthy Diet

INTERVENTIONS:
Behavioral: Healthy Diet — Receive counseling to meet guidelines for healthy dietary patterns
  Arms: Healthy Diet

SUMMARY:
The overall aim of the present research program is to determine how a healthy whole-diet approach impacts on cardiometabolic health in adults. With its interdisciplinary approach, the study depicts mechanisms behind disease progression and the impact of healthy dietary patterns on changes in markers of low-grade systemic inflammation together with the exploration of knowledge and attitudes about healthy diets. The study has a preventive character as it targets older adults (65+) without manifest disease.

DETAILED DESCRIPTION:
This two arm randomized-controlled study includes the following groups: Controls and Healthy Diet group.

The study will particularly address the following aspects:

* determine food literacy, perceived attitudes and barriers for the adoption of new dietary habits incorporating increased fruit and vegetable intake in adults.
* explore the effects of a randomized controlled intervention promoting healthy dietary patterns (increased intakes of fruit and vegetable, whole-grain, nuts and low fat dairy products and replacing saturated with unsaturated fats and decreased red meat and salt consumption) for a period of 4 months on components of the metabolic syndrome, a large panel of pro- and anti-inflammatory biomarkers and metabolomic profile in adults.
* assess the long-term adherence to healthy dietary patterns in adults.
* provide support for behavioural change and evaluate participants' perception of this support.

ELIGIBILITY:
Inclusion Criteria:

* 65-70 years
* not meeting 5 servings of fruit and vegetable per day
* Waist circumference >80 cm (female) and >88 (male)

Exclusion Criteria:

* Movement disability
* Diabetes, cardiovascular disease, lung disease, overt disease

Ages: 65 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose | Before and after 16 weeks
  Blood glucose (mmol/L) assessed using chemistry kits from Ortho-Clinical Diagnostics on a Vitros-5.1 analyzer platform (Clinical Diagnostics, Raritan, NJ, United States)
Change in plasma triglycerides | Before and after 16 weeks
  Plasma triglycerides (mmol/L) : assessed using chemistry kits from Ortho-Clinical Diagnostics on a Vitros-5.1 analyzer platform (Clinical Diagnostics, Raritan, NJ, United States)
Change in high-density lipoprotein cholesterol | Before and after 16 weeks
  high-density lipoprotein cholesterol (mmol/L) : assessed using chemistry kits from Ortho-Clinical Diagnostics on a Vitros-5.1 analyzer platform (Clinical Diagnostics, Raritan, NJ, United States)
Change in waist circumference | Before and after 16 weeks
  waist circumference (cm) assessed by a steel tape
Change in diastolic and systolic blood pressure (mmHg) | Before and after 16 weeks
  diastolic and systolic blood pressure (mmHg) assessed using a manual sphygmomanometer
Change in intake of fruit and vegetable | Before and after 16 weeks
  - Fruit and vegetable intake assessed on a 7 scale-item where the lowest value of 1, indicates an intake less than 1 per month, and 7 an intake of at least 5 servings /day.

CONTACTS AND LOCATIONS:
Overall Officials: Fawzi Kadi, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data on participant characteristics and main study outcomes will be made available on reasonable request when the results are published.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data are available once the results are published.
Access Criteria: Controlled access will be applied as follows:
  For secondary users (researchers):
  * registration and data use agreement are required
  * review of secondary users' qualifications, research proposals and data analysis plans.
  For trial participants:
  - Own individual data will be available upon request.

REFERENCES:
- [Derived] Bergens O, Veen J, Montiel-Rojas D, Edholm P, Kadi F, Nilsson A. Impact of healthy diet and physical activity on metabolic health in men and women: Study Protocol Clinical Trial (SPIRIT Compliant). Medicine (Baltimore). 2020 Apr;99(16):e19584. doi: 10.1097/MD.0000000000019584. PMID 32311926